CLINICAL TRIAL: NCT03147495
Title: Research on the Association Between the Inclination of the Proximal Tibiofibular Joint Surface and Medial Compartment Knee Osteoarthritis
Brief Title: The Inclination of the Proximal Tibiofibular Joint Surface and Medial Compartment Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: 113th Hospital of Chinese People's Liberation Army (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Other Study IDs: 113YY-LUNLI-2017005
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the study group: The participants with medial compartment knee osteoarthritis and without lateral compartment knee osteoarthritis according to the Ahlbäck classification.
  Interventions: Diagnostic Test: Standing anteroposterior knee radiographs and special proximal tibiofibular joint radiograph.
- the control group: The healthy volunteers without knee osteoarthritis according to the American College of Rheumatology criteria for the classification and reporting of OA of the knee joint. Radiographic evidence of the knee with Ahlbäck classification grade 0.
  Interventions: Diagnostic Test: Standing anteroposterior knee radiographs and special proximal tibiofibular joint radiograph.

INTERVENTIONS:
Diagnostic Test: Standing anteroposterior knee radiographs and special proximal tibiofibular joint radiograph. — Standing anteroposterior knee radiographs and special proximal tibiofibular joint radiographs will be taken for the participants in both groups. The standing anteroposterior knee radiographs will be obtained with the knee extended. The proximal tibiofibular joint radiographs will be acquired with the knee of the participants in approximately 45°-60° of internal rotation.

SUMMARY:
This study aims to research on the association between the inclination of the proximal tibiofibular joint surface and medial compartment knee osteoarthritis. The proximal tibiofibular joint radiographs of the participants will be taken. The angle of inclination of the proximal tibiofibular joint surface in two groups will be compared.

DETAILED DESCRIPTION:
The nonuniform settlement of the tibial plateau has been introduced to explain the development of knee varus and medial compartment knee osteoarthritis. It is believed that the lateral support of the fibula to the tibial plateau leads to the nonuniform settlement and degeneration of the plateau bilaterally.

Bone mass decreases as part of the normal aging process. Varying degrees of settlement of bone mass exist in the load-bearing joints, such as the knees, hips, ankles, and spine. In the proximal tibia, the lateral support of the fibula to the lateral tibial plateau routinely leads to nonuniform settlement, which is more severe in the medial plateau than in the lateral plateau. The slope of the tibial plateau arising from nonuniform settlement results in a transverse shearing force, with the femoral condyle shifting medially during walking and sports. Furthermore, side-slip aggravates the nonuniform settlement of the tibial plateau, especially in the medial plateau. Accordingly, a cycle of increasing the load distribution in the medial compartment and nonuniform settlement occurs. This results in the load from the normal distribution shifting farther medially to the medial plateau and consequently leads to knee varus, aggravating the progression of medial compartment knee osteoarthritis.

However, the angle of inclination of the proximal tibiofibular joint surface in different individuals varied widely. The angle of inclination of the proximal tibiofibular joint may affect the nonuniform settlement of the bilateral tibial plateau.

This study aims to research on the association between the inclination of the proximal tibiofibular joint surface and medial compartment knee osteoarthritis. A sample size power analysis was conducted before the study, which revealed that a minimum of 39 subjects per group was needed to achieve statistical significance with two-sided α=0.05 and 1-ß=0.80 and an assumed mean differences between two groups = 65% of the standard deviation.

Participants will be recruited from the outpatient clinic of No.113 Hospital of Chinese People's Liberation Army, as well as advertising flyers within the clinic. Firstly, patients of the study group will be recruited. It is hoped that the number of males will be equal to the number of females. Then the controls will be recruited and matched for age (within 5 years) and sex to the cases.

Standing anteroposterior knee radiographs and special PTFJ radiographs will be taken for the participants in both groups. The standing anteroposterior knee radiographs will be obtained with the knee extended. The PTFJ radiographs will be acquired with the knee of the participants in approximately 45°-60° of internal rotation.

On weight bearing anteroposterior radiographs of knee, osteoarthritis will be graded by using the Ahlbäck grading scale, and femorotibial angle will be measured. The Ahlbäck classification Stage 0: No radiographic sign of arthritis. Stage I: Narrowing of the joint space (JSN) (with or without subchondral sclerosis). JSN is defined by a space inferior to 3 mm, or inferior to the half of the space in the other compartment (or in the homologous compartment of the other knee). Stage II: Obliteration of the joint space; Stage III: Bone defect/loss <5 mm. Stage IV: Bone defect/loss between 5 and 10 mm. Stage V: Bone defect/loss >10 mm, often with subluxation and arthritis of the other compartment.

For the PTFJ radiographs, the degenerative joint disease of the PTFJ will be staged with the Kellgren-Lawrence staging system, and the fibular inclination angle (FIA) and the tibial inclination angle (TIA) of the PTFJ surface to the longitudinal axis of both fibula and tibia will be measured separately. The Kellgren-Lawrence Grade 0: No X-ray changes of osteoarthritis. Grade I: Formation of osteophytes on the joint margins, in the knee joint, on the tibial spine. Grade II: Grade I + thinning of joint cartilage associated with sclerosis of subchondral bone. Grade III: Grade I + II + subchondral cysts. Grade IV: Grade I + II + III + deformation of the bone ends.

Demographics, laterality of included knees and FTA, the inclination angle of the proximal tibiofibular joint surface and the grade of the proximal tibiofibular joint degeneration in two groups will be evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic knee osteoarthritis according to the American College of Rheumatology criteria for the classification and reporting of OA of the knee joint,
* predominance of self-reported pain over the medial aspect of the knee,
* radiographic evidence of medial compartment knee osteoarthritis with an Ahlbäck score of grade I or greater,
* and radiographic evidence of lateral compartment with Ahlbäck classification grade 0.

Exclusion Criteria:

* any previous surgery or severe trauma in the affected limb.
* inflammatory joint disease or tumors in the affected limb.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The outpatient clinic of No.113 Hospital of Chinese People's Liberation Army
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2020-09-13 (Actual); Study Completion 2020-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qingsheng Zhu, MD, Study Director — Department of orthopaedics, Xijing hospital, Fourth Military Medical University, Xi'an, China
Locations (1):
- Orthopaedics clinic, No.113 Hospital of Chinese People's Liberation Army, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were enrolled at the outpatient clinic of our hospital. The patients with medial compartment knee osteoarthritis were enrolled at first. The anticipated number of patients was 40, and the female-to-male ratio was expected to be 1:1. Then, the participants of the control group were enrolled and matched for sex and age (within 5 years) to the patients. The control-to-patient ratio was 1:1.
Groups:
- the Study Group: The participants with medial compartment knee osteoarthritis and without lateral compartment knee osteoarthritis according to the Ahlbäck classification.
  no intervention: The proximal tibiofibular joint radiographs will be taken for the participants in both groups.
- the Control Group: The healthy volunteers without knee osteoarthritis according to the American College of Rheumatology criteria for the classification and reporting of OA of the knee joint. Radiographic evidence of the knee with Ahlbäck classification grade 0.
  no intervention: The proximal tibiofibular joint radiographs will be taken for the participants in both groups.
Period: Overall Study
Arm/Group | the Study Group | the Control Group
Started | 40 | 46
Completed | 40 | 40
Not Completed | 0 | 6
Not completed — Physician Decision | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | the Study Group | the Control Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.08 (6.84) | 61.10 (7.60) | 62.59 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 20 | 20 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 40 | 40 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 40 | 40 | 80
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26.26 (3.72) | 24.84 (2.78) | 25.55 (3.34)
Laterality of knee [Count of Participants; unit: Participants] — The laterality of knee was choosed by the participant or investigators.
  Participants
    Right knee | 24 | 20 | 44
    Left knee | 16 | 20 | 36

OUTCOME MEASURES:

1. Primary Outcome: The Fibular Inclination Angle of the Proximal Tibiofibular Joint Surface
Description: The fibular inclination angle of the proximal tibiofibular joint surface to the longitudinal axes of both tibia and fibula
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | the Study Group | the Control Group
Number analyzed (Participants) | 40 | 40
degrees | 26.82 (7.97) | 31.99 (7.92)

2. Primary Outcome: The Tibial Inclination Angle of the Proximal Tibiofibular Joint Surface
Description: The tibial inclination angle of the proximal tibiofibular joint surface to the longitudinal axes of both tibia and fibula
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | the Study Group | the Control Group
Number analyzed (Participants) | 40 | 40
degrees | 26.91 (7.30) | 33.44 (6.85)

3. Secondary Outcome: Grade of the Proximal Tibiofibular Joint Degeneration
Description: Arthritic grades of the proximal tibiofibular joint were staged with Kellgren-Lawrence staging system.
  The Kellgren-Lawrence Grade 0: No X-ray changes of osteoarthritis. Grade I: Formation of osteophytes on the joint margins, in the knee joint, on the tibial spine. Grade II: Grade I + thinning of joint cartilage associated with sclerosis of subchondral bone. Grade III: Grade I + II + subchondral cysts. Grade IV: Grade I + II + III + deformation of the bone ends. The higher the Kellgren-Lawrence Grade is, the more severe the proximal tibiofibular joint degeneration.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | the Study Group | the Control Group
Number analyzed (Participants) | 40 | 40
Participants
  grades 0 | 20 | 30
  grade Ⅰ | 14 | 8
  grade Ⅱ | 6 | 2
  grade Ⅲ | 0 | 0
  grade Ⅳ | 0 | 0

4. Secondary Outcome: The Femorotibial Angle
Description: The lateral angle between the femoral axis and the tibial axis measured on an weight bearing anteroposterior radiograph of knee
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | the Study Group | the Control Group
Number analyzed (Participants) | 40 | 40
degrees | 179.34 (3.60) | 174.37 (2.65)

5. Secondary Outcome: The Fibular PTFJ Types
Description: The horizontal fibular PTFJ type was defined as the fibular inclination angle ≤ 20°, and the oblique fibular PTFJ type was defined as the fibular inclination angle > 20°.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | the Study Group | the Control Group
Number analyzed (Participants) | 40 | 40
Participants
  horizontal type | 9 | 3
  oblique type | 31 | 37

6. Secondary Outcome: The Tibial PTFJ Types
Description: The horizontal tibial PTFJ type was defined as the tibial inclination angle ≤ 20°, and the oblique tibial PTFJ type was defined as the fibular inclination angle > 20°.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | the Study Group | the Control Group
Number analyzed (Participants) | 40 | 40
Participants
  horizontal type | 8 | 2
  oblique type | 32 | 38

ADVERSE EVENTS:
Time Frame: half an hour
Arm/Group | the Study Group | the Control Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/46
Other Adverse Events (participants affected / at risk) | 0/40 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT03147495/Prot_SAP_000.pdf